CLINICAL TRIAL: NCT04839315
Title: Immunological Consequences of COVID-19 Vaccination in Patients With Rheumatic Diseases
Brief Title: COVID-19 Vaccination in Rheumatic Disease Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hu Zeng, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-000501
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Systemic Lupus Erythematosus; Sjogren's Syndrome; Inflammatory Myositis; Psoriatic Arthritis; Gout; Ankylosing Spondylitis; Arthritis of Multiple Sites Associated With Inflammatory Bowel Disease (Diagnosis); Osteoarthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sjogren's Syndrome; Arthritis, Psoriatic; Gout; Spondylitis, Ankylosing; Disease; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA COVID19 vaccines (Other): mRNA-based COVID19 vaccines
  Interventions: Biological: mRNA COVD19 vaccine

INTERVENTIONS:
Biological: mRNA COVD19 vaccine — Subjects will receive two doses of mRNA based COVID19 vaccines.

SUMMARY:
The research is being done to study the immune responses to COVID-19 vaccination in patients with rheumatic diseases.

DETAILED DESCRIPTION:
Because patients treated with immunosuppressive agents have been excluded from initial clinical trials, and most patients with rheumatic diseases are taking immunosuppressants, the immune responses towards the mRNA COVID19 vaccines in these patients remains unknown. The goal is to study the immune response to COVID-19 vaccination in patients with rheumatic diseases. Blood samples collected before and longitudinally after mRNA-based COVID-19 vaccination (i.e., Pfizer and Moderna vaccines) will enable detailed immunological investigation of the interaction between COVID-19 vaccination and rheumatic diseases. These efforts will provide novel insights into the COVID-19 vaccine response in patients with rheumatic diseases, and eventually would inform clinical management to improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologist confirmed diagnosis of one of the following diagnoses:
* Systemic lupus erythematosus;
* Sjogren syndrome;
* Inflammatory myositis;
* Psoriatic arthritis;
* Osteoarthritis;
* Gout;
* Ankylosing spondylitis;
* IBD-related arthritis.

Exclusion Criteria:

* Active infection or untreated malignancy (other than skin cancer) at enrollment.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Humoral responses towards mRNA COVID-19 vaccines | 2 weeks to 6 months after second dose of vaccine
  We aim to examine SARS-Cov2 specific antibody, and autoantibody generation

SECONDARY OUTCOMES:
Cellular immune responses towards mRNA COVID-19 vaccines | 2 weeks to 6 months after second dose of vaccine
  measurement of immune cell distributions, type I interferon activity, and SARS-Cov2 specific T cell responses

CONTACTS AND LOCATIONS:
Overall Officials: Hu Zeng, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials